CLINICAL TRIAL: NCT05599906
Title: Effects of Inpatient Rehabilitation Measures in Long-COVID-19 Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paracelsus Harz Clinic Bad Suderode. (Other)
Responsible Party: Sponsor
Other Study IDs: 96/21
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-10

CONDITIONS: Long COVID
Keywords: long covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: questionnaires — Completion of 3 questionnaires (HADS; SF-12; FAS) at the beginning and end of the rehabilitation and after 3 months

SUMMARY:
The aim of the present study is to answer the question of whether a rehabilitation measure has a positive effect on fatigue symptoms, physical performance, and the physical and psychological well-being of the patients. In particular, the fatigue that occurs in most of all patients is of interest here. In order to make this measurable, the FAS questionnaire plays a special role, which should be completed by all 100 patients upon inclusion in the study and upon discharge from the rehabilitation clinic. In addition, the HADS-D questionnaire (Hospital Anxiety and Depression Scale) for self-assessment of depressive symptoms and anxiety symptoms and the SF-12 questionnaire (Short Form Health Survey) are used as a screening tool to assess health-related quality of life.

For the clinical examination of physical performance, the six-minute walk test, a body plethysmography and a long-term ECG are performed on recruited patients on admission and before discharge. In a three-month follow-up, all recruited patients should receive an FAS, HADS-D and SF-12 questionnaire to fill out. Some of these will also be called back to the clinic to check the development of lung function or performance, defined on the basis of VO2max, and will undergo an additional spiroergometric examination.

Thus, the effectiveness and effectiveness of the rehabilitation measures in patients under long-COVID is checked.

DETAILED DESCRIPTION:
The study is a prospective, monocentric cohort study in which patients with the main diagnosis of long-COVID syndrome from the Paracelsus Harz Clinic, Bad Suderode, are included and followed up over a period of three months.

The study population consists of patients from the rehabilitation clinic Paracelsus-Harz-Klinik Bad Suderode. It is planned to enroll 100 patients, all of whom will be included in a three-month follow-up. Within this follow-up, 20 of the 100 patients will be selected to be re-examined in the clinic three months later. For this purpose, patients are selected who live within a maximum distance of 50km from the Paracelsus Harz Clinic and who are able to reach the clinic three months after completion of the rehabilitation measure.

After receiving the vote of the Ethics Committee of the Medical Association of the State of Saxony-Anhalt (Bad Suderode) and the written consent of the patients, socio-demographic information and questions are documented according to the standard of the rehabilitation clinic. All relevant baseline parameters (age, gender, BMI, drug treatment, etc.) are also documented. In order to obtain the essential values for the evaluation of the physical and psychological condition of the patients, all patients receive an FAS questionnaire, a HADS-D and an SF-12 questionnaire upon inclusion and at the end of the rehabilitation stay. Furthermore, after admission and before discharge, a six-minute walk test, a lung function test using body plethysmography and a long-term ECG for cardiological observation are carried out.

After the patients have left the clinic, 80 of the recruited patients will be contacted by post three months later in order to fill out the previously known questionnaires again. The Fatigue Questionnaire (FAS Questionnaire) is of particular interest for checking the physical and psychological development after completion of the rehabilitation treatment. In addition, the patients should again receive the HADS-D and SF-12 questionnaires to check their mental and physical well-being. If the patients cannot be reached, an attempt is made to obtain follow-up information by telephone, relatives or general practitioners. The remaining 20 patients will be referred to the clinic again as part of the three-month follow-up so that the development of lung function and performance, measured using VO2max, can be checked in the form of spiroergometry. During their stay, they also receive the FAS questionnaire, the HADS-D and the SF-12 questionnaire to fill out

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years, written consent; inpatient stay in the participating rehabilitation clinic

Exclusion Criteria:

* lack of consent, Illnesses or functional disorders which, in the opinion of the investigator, exclude participation in this clinical trial (dementia, psychotic disorders)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with long/post-covid
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Course of fatigue symptoms measured with the FAS score | Day one
  Analysis of the questionnaires
Course of fatigue symptoms measured with the FAS score | after 3 weeks
  Analysis of the questionnaires
Course of fatigue symptoms measured with the FAS score | after 3 Months
  Analysis of the questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Harzklinik Bad Suderode GmbH, Quedlinburg, Germany